CLINICAL TRIAL: NCT03193281
Title: KISS Study: A Phase II Study of Dasatinib Followed by Imatinib in Newly Diagnosed, Previously Untreated Patients With Chronic Phase CML
Brief Title: KISS Study: Kinase Inhibition With Sprycel Start up
Acronym: KISS
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Auckland, New Zealand (Other)
Collaborators: Leukaemia & Blood Cancer New Zealand (Unknown)
Responsible Party: Principal Investigator, Peter Browett, Professor, University of Auckland, New Zealand
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTNZ-2012-08
Record Dates: First submitted 2017-06-15; First posted 2017-06-20 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Chronic Myeloid Leukemia
Keywords: Dasatinib; Imatinib
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — Dasatinib; Imatinib Mesylate

STUDY DESIGN:
Intervention Model Description: A Phase II, multicentre, open-label, prospective non-randomised study of treatment modification in response to maintenance of MR3.0 at 12 months.
  Molecular response will be measured 3 monthly. Patients who achieve MR3.0 by 12 months, with a confirmed response at 13 months on treatment, will switch treatment to imatinib. Those patients who do not achieve this confirmed response will remain on dasatinib.
  For patients who achieve confirmed MR3.0 by 13 months we define two study stages. Stage 1 is the first 12 months after recruitment (i.e. before the possible switch to imatinib) and Stage 2 includes the months 13 - 37.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Dasatinib (Other): All patients will begin the study on dasatinib treatment (Sprycel® 100mg once daily oral administration). Those who reach MR3.0 at 12 months (end of Study Stage 1) and achieve a confirmed result at 13 months, will switch to imatinib treatment (Imatinib-AFT 400mg once daily oral administration) for the next 24 months (Study Stage 2).
  Patients who do not achieve a confirmed MR3.0 result at 13 months will not be eligible to switch to imatinib treatment and will remain on dasatinib treatment, as per Study Stage 1.
  Patients will be assessed on a 3-monthly basis throughout the study. Those who discontinue dasatinib treatment during the study for reasons other than the planned treatment switch to imatinib at 13 months, will also be followed up every 3 months.
  Interventions: Drug: Dasatinib; Drug: Imatinib

INTERVENTIONS:
Drug: Dasatinib — In order to test the study hypothesis patients need to stay on dasatinib (Sprycel) treatment for the first 12 months of the study (Stage 1).
  Patients who do not reach MR3.0 at 12 months will remain on dasatinib treatment.
  Other Names: Sprycel
Drug: Imatinib — Patients who reach MR3.0 at 12 months (and the result is confirmed at 13 months) will switch to imatinib (Imatinib-AFT) treatment.
  Other Names: Imatinib-AFT

SUMMARY:
Chronic myeloid leukaemia (CML) is due to a chromosomal abnormality in white blood cells which results in abnormal multiplication. CML in its earlier, slower growing chronic phase (CP) is well controlled by the tyrosine kinase inhibitor (TKI) drug imatinib, which targets the consequences of the chromosomal abnormality, inducing a response and subsequent remission (as measured using molecular techniques on patient blood or bone marrow samples in the lab). Dasatinib, a newer TKI drug, similar in design to imatinib, gives a more rapid molecular response, however the long term side-effects are less known than imatinib.

This study will investigate the efficacy and safety of a treatment plan for patients with newly diagnosed CML-CP, where dasatinib will be used to more rapidly induce a molecular response (MR3.0) within 12 months, after which imatinib will be used to maintain the CML in that remission. It is hypothesised that imatinib is safe and effective in maintaining MR3.0 in patients with CML who achieve MR3.0 at 12 months following initial induction therapy with dasatinib.

DETAILED DESCRIPTION:
The KISS Study is a Phase II, multicentre, open-label, prospective non-randomised study of treatment modification in response to maintenance of MR3.0 at 12 months. Patients must be newly diagnosed with chronic phase CML (CML-CP) (<3 months) and previously untreated with the exception of hydroxyurea.

Patients will be recruited from hospital haematology clinics. The majority of patients will have been referred to a haematologist due to suspected CML. Written informed consent will be ensured before any study-specific procedures are undertaken or study data collected, however the majority of assessments carried out for this study are based on standard of care.

Patients' eligibility will be determined by the usual procedures carried out for CML diagnosis. Results from both diagnostic procedures and confirmatory screening procedures will constitute baseline data. Once a patient has had their eligibility confirmed and has signed informed consent, they will be enrolled into the trial.

The trial consists of two stages:

Stage 1: The first 12 months after recruitment (before the possible switch to imatinib).

Stage 2: Months 13 - 37.

The following measurements/data will be recorded throughout the trial at protocol specified time points:

* Haematology and biochemistry.
* PB Q-PCR for BCR-ABL1.
* Chest x-ray, ECG, ECHO.
* Medical assessment including physical exam, ECOG performance, weight, vital signs, assessment of extra medullary disease (liver, lymph nodes and spleen), spleen measurement below left costal margin, adverse events and concomitant medications.
* Haematological and molecular response assessments.
* Treatment adherence assessment.
* Patient questionnaire (MDASI-CML).

All patients will commence dasatinib (Sprycel®) 100 mg daily. Molecular monitoring of blood BCR-ABL1 transcripts to measure molecular response will occur 3 monthly by Q-PCR as per standard of care procedures. Patients who achieve a BCR-ABL1 level of ≤ 0.1% (MR3.0) by 12 months on treatment will switch treatment to imatinib 400 mg daily if MR3.0 is confirmed at 13 months (and they give their consent to switch). Those patients who do not achieve MR3.0 at 12 months or MR3.0 is not confirmed at 13 months, will remain on dasatinib. Patients with confirmed MR3.0 who choose not to switch to imatinib will continue on dasatinib. Patients that are intolerant of dasatinib in the first 12 months, those that switch to imatinib at 12 months and then lose MR3.0 or those intolerant of imatinib will be treated off study.

ELIGIBILITY:
INCLUSION CRITERIA:

1. Male or female patients ≥ 18 years of age.
2. ECOG performance status score of 0-2.
3. Patients must have all of the following:

   1. Be enrolled within 3 months of initial diagnosis of CML-CP (date of initial diagnosis is the date of first cytogenetic analysis).
   2. Cytogenetic or molecular confirmation of Ph+ or variants of (9;22) translocations.

      patients may have secondary chromosomal abnormalities in addition to the Ph+.
   3. Documented chronic phase CML as defined by:

      * < 15% blasts in peripheral blood and bone marrow.
      * < 30% blasts plus promyelocytes in peripheral blood and bone marrow.
      * < 20% basophils in peripheral blood.
      * ≥ 100 x 109/L platelets (unless considered related to hydroxyurea).
      * no evidence of extramedullary leukaemic involvement, with the exception of hepatosplenomegaly.
   4. BCR-ABL1 transcript that can be monitored by Q-PCR.
   5. Baseline full blood count (within 14 days of enrolment) remains consistent with chronic phase CML criteria.
4. Voluntary written informed consent.

EXCLUSION CRITERIA:

1. Any prior treatment for CML with other than hydroxyurea.
2. Patients with the following laboratory values:

   1. serum bilirubin > 2.0 x the institutional upper limit of the normal range (ULN).
   2. ALT > 2.0 x the institutional upper limit of the normal range (ULN).
   3. creatinine > 2.0 x the institutional upper limit of the normal range (ULN).
   4. International normalised ratio (INR) or partial thromboplastin time (PTT) > 1.5 x ULN, with the exception of patients on treatment with oral anticoagulants.
3. Patients with uncontrolled medical disease such as diabetes mellitus, thyroid dysfunction, neuropsychiatric disorders or infection.
4. Patients with:

   1. Grade 3/4 cardiac problems as defined by the New York Heart Association Criteria.
   2. Uncontrolled hypertension.
   3. Grade 3/4 respiratory dysfunction.
   4. Past or current history of pleural effusions or pulmonary arterial hypertension.
5. Patients with known positivity for human immunodeficiency virus (HIV); baseline testing for HIV is not required.
6. Patients who have undergone major surgery within 4 weeks of study Day 0, or who have not recovered from prior major surgery.
7. Patients who are:

   1. pregnant.
   2. breast feeding.
   3. of childbearing potential without a negative pregnancy test on/prior to Day 0.
   4. male or female of childbearing potential unwilling to use barrier contraceptive precautions throughout the trial (postmenopausal women must be amenorrhoeic for at least 12 months to be considered of non-childbearing potential).
8. Patients with another uncontrolled malignancy with the exception of basal cell skin carcinoma or cervical carcinoma in situ.
9. Patients with positivity for hepatitis B antigen and / or hepatitis B core antibody (unless receiving prophylactic therapy with lamivudine or more potent agent)
10. Patients with a history of non-compliance to medical regimens or who are considered potentially unreliable.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2017-07-17 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
To estimate the proportion of patients who remain in MR3.0 for the duration of 2 years following a change of therapy from dasatinib to imatinib at 13 months. | 2 years

SECONDARY OUTCOMES:
To estimate progression free survival (PFS), failure free survival (FFS) and overall survival (OS) for patients that switch to imatinib at 13 months. | 3 years
To estimate the proportion of patients who regain MR3.0 on dasatinib or another TKI therapy after having a confirmed loss of MR3.0 on imatinib, for patients that switch to imatinib at 13 months. | 3 years
To estimate time to MR3.0, MR4.5 and MR5.0 for patients that switch to imatinib at 13 months. | 3 years
To describe adverse event profiles on Stage 1 and Stage 2 of the study and overall for patients that switch to imatinib at 13 months. | 3 years
To describe the quality of life on Stage 1 and Stage 2 of the study and overall for those that switch to imatinib at 13 months. | 3 years

OTHER OUTCOMES:
To estimate PFS, FFS and OS for the following groups: 1) the entire cohort 2) patients not eligible to switch to imatinib at 13 months 3) patients that are eligible but do not switch. | 3 years
To estimate time to MR3.0, MR4.5 and MR5.0 for the following groups: 1) the entire cohort 2) patients not eligible to switch to imatinib at 13 months 3) patients that are eligible but do not switch. | 3 years
To describe adverse event profiles on each stage of study therapy for the following groups: 1) the entire cohort 2) patients not eligible to switch to imatinib at 13 months 3) patients that are eligible but do not switch. | 3 years
To describe the quality of life on each stage of study therapy for the following groups: 1) the entire cohort 2) patients not eligible to switch to imatinib at 13 months 3) patients that are eligible but do not switch. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Peter Browett, MBChB, Principal Investigator — University of Auckland, New Zealand
Locations (9):
- New Zealand (9):
  - Auckland City Hospital, Auckland
  - Middlemore Hospital, Auckland
  - Christchurch Hospital, Christchurch
  - Dunedin Hospital, Dunedin
  - Waikato Hospital, Hamilton
  - Taranaki Base Hospital, New Plymouth
  - Palmerston North Hospital, Palmerston North
  - North Shore Hospital, Takapuna
  - Wellington Hospital, Wellington

IPD SHARING:
Plan to Share IPD: No